CLINICAL TRIAL: NCT00256230
Title: Evaluation of Disulfiram in Patients With Metastatic Melanoma and at Least One Prior Systemic Therapy, Phase I/II
Brief Title: Disulfiram in Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: John P. Fruehauf (Other)
Responsible Party: Sponsor-Investigator, John P. Fruehauf, Dr. John P. Fruehauf, University of California, Irvine
Organization: University of California, Irvine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCI 01-01; 2001-2038 (Other: University of California, Irvine)
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — Disulfiram

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Disulfiram (Experimental)
  Interventions: Drug: Disulfiram (DSF)

INTERVENTIONS:
Drug: Disulfiram (DSF) — DSF pills at 250 mg will be given orally, two times a day. If this dose is tolerated, the dose will be escalated until the maximum tolerated dose is reached. Treatment will continue every day for 3 months or longer unless the disease gets worse, the side effects are too dangerous for the subject, or the subject decides to discontinue treatment.
  Other Names: bis(diethylthiocarbamoyl) disulfide

SUMMARY:
Melanoma remains a malignancy that is largely resistant to chemotherapy. Metastatic disease responds poorly to the treatments used today with only 2 out of 30 drugs tested, DTIC and nitrosoureas, showing response rates greater than 10%, and complete responses are rare. DTIC-based regimen has been recognized as a standard chemotherapy for advanced melanoma, and temozolomide demonstrated efficacy equal to that of DTIC and is an oral alternative agent that also crosses the blood brain barrier. Randomized phase III trials have shown no survival benefit of adding other agents (cisplatin, BCNU, and tamoxifen). Biochemotherapy is being developed extensively with moderate improvement in the responsive rate (approximately 50%) and is under evaluation in randomized trial to identify whether there is survival benefit to this strategy, compared with chemotherapy alone. Recently, a randomized phase III study comparing chemotherapy (cisplatin, dacarbazine, and tamoxifen) with biochemotherapy (the same chemotherapy regimen plus high-dose IL-2 and interferon alfa) have shown 44% response rate for biochemotherapy vs. 27% for chemotherapy. However, the tendency toward an increased response rate in patients who received biochemotherapy did not translate into an increase in overall survival, and there was, in fact, a trend for a survival advantage in patients receiving chemotherapy alone (median survival: 10.7 vs 15.8 months). New agents (or combinations) need to be developed for this refractory malignancy.

The purpose of this study is to determine the response rate and evaluate the toxicity of disulfiram (DSF) in the treatment of Stage IV melanoma.

The advantages of using DSF in this phase I/II trial are the following:

* DSF has been used as a drug for many years for the treatment of alcoholism. Its mechanism, pharmacokinetics, toxicity/tolerable dose are well known, and this drug is relatively non-toxic by itself at therapeutic dose. Doses of greater than 3000mg/m2 can cause reversible confusion.
* DSF can be taken orally; therefore, it is convenient to administer.
* DSF can penetrate the blood-brain barrier (unlike dacarbazine and many other chemotherapy agents); therefore, it might have an active effect on CNS metastasis.

This study is designed to include women and minorities, but is not designed to measure differences of intervention effect.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be between the ages of 18 and 80.
* Patient must have pathologically proven and surgically incurable malignant melanoma, which is Stage IV.
* Patient must have bidimensionally measurable disease. All measurable lesions must be assessed (by physical examination, CT scan, radionuclide scan or plain X-ray) within 28 days prior to registration. Non-measurable sites must be assessed within 42 days prior to registration. The patient's disease status must be completely assessed and reported.
* All patients must undergo a CT of abdomen and chest within 28 days prior to registration.
* All patients must undergo either a CT or MRI of the brain within 28 days of registration. Patients with or without brain metastasis are both recruited for this protocol.
* Patients must have received at least one prior systemic therapy (chemotherapy, biologic/immunotherapy, or a combination regimen) for metastatic disease. Prior systemic therapy must have been completed at least 28 days before registration.
* Patients may have received prior biologic or immunotherapy given in an adjuvant fashion. Prior adjuvant therapy must have been completed at least 28 days prior to registration
* Patients may have received prior radiation therapy. If all known sites of disease have been previously radiated, there must be objective evidence of progression for the patient to be eligible. Radiation therapy must have been completed at least 28 days before registration.
* Patients may have received prior surgery. Prior surgery must have been completed at least 28 days before registration.
* Performance status must be 0-2 according to Zubrod Criteria.
* If day 28 or 42 falls on a weekend or holiday, the limit may be extended to the next working day.
* Patients must be informed of the investigational nature of this study and sign and give written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* Patients with severe myocardial disease or coronary occlusion, psychoses, and hypersensitivity to disulfiram or other thiuram derivatives used in pesticides and rubber vulcanization are excluded from the study.
* Patients who cannot abstain from alcohol intake during the entire duration of this protocol are not qualified for this study.
* Patients requiring ongoing therapy with other investigational drugs are excluded.
* Pregnant or nursing women are not eligible to participate in this trial because the safe use of this drug in pregnancy has not been established.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2002-01; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Determine response rate | Every 8 weeks during therapy
  Complete response (CR)-Complete disappearance of all measurable and evaluable disease. No disease related symptoms. No evidence of non-evaluable disease, including normalization of markers and other abnormal lab values. Partial response (PR)-Applies only to patients with at least one measurable lesion. Greater than or equal to 50% decrease under baseline in the sum of products of perpendicular diameters of all measurable lesions. No progression of evaluable disease. For both CR and PR, no new lesions. All assessments use the same techniques as baseline.

SECONDARY OUTCOMES:
Evaluate the toxicity of disulfiram administration | Lab tests-Weeks 2, 4, 8, 12, 16, 20 and 24; X-rays/scans-Every 8 weeks
  Accelerated titration designs are used for the maximum tolerated dose.
  Patients will remain at one dose level for one week before escalated to the next higher dose level, providing that no grade II or III toxicity occurs.
  Phase II is to use the maximum tolerated dose of DSF (as described above) to determine the response rate. Evaluation of toxicities will be continued. Dose reduction (switch to the next lower dose) will be carried out if patient develops grade III/IV toxicities, and this dose reduction applies to both phase I and phase II.

CONTACTS AND LOCATIONS:
Overall Officials: John Fruehauf, MD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, Orange, California, United States